CLINICAL TRIAL: NCT04897490
Title: Real World Evidence of First Line Treatment With Arsenic Trioxide Plus All Trans Retinoic Acid in Adult Patients With Acute Promyelocytic Leukemia
Brief Title: RWE of 1st Line Treatment With ATO/ATRA for Adult APL
Status: Recruiting | Type: Observational
Sponsor: Grupo Argentino de Tratamiento de la Leucemia Aguda (Other)
Responsible Party: Sponsor
Other Study IDs: GATLA 11-LPA-20
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Promyelocytic Leukemia, Adult Acute
Keywords: Acute Promyelocytic Leukemia; ATRA; ATO; IDA
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult APL in first line: Patients >/= 18 years old with recent diagnosis of acute promyelocytic leukemia who receive treatment with ATO/ATRA according to our local guidelines. HR patients will receive 2-3 additional doses of idarubicin.
  Interventions: Other: Evaluation of first line treatment with ATO/ATRA outcome

INTERVENTIONS:
Other: Evaluation of first line treatment with ATO/ATRA outcome — Evaluation of first line treatment with ATO/ATRA outcome (o event free survival and overall survival and toxicity) in adult patients with APL.

SUMMARY:
This is a multicenter, observational real world clinical trial with prospective follow up that will evaluate the treatment outcome of acute promyelocytic leukemia (APL) patients in the first line with arsenic trioxide and all trans retinoic acid (ATO/ATRA) based regimens in Argentina.

DETAILED DESCRIPTION:
The purpose of this trial is to gather real world evidence of the characteristics of APL patients in Argentina who receive ATO/ATRA based treatment in first line following our national guidelines. The study primary endpoint is to evaluate event free survival and overall survival of patients diagnosed with APL and treated in first line with ATO/ATRA or ATO/ATRA/Idarubicin (IDA) depending on risk category. Secondary endpoints are complete molecular response (CMR) rate, toxicity, early mortality and prognostic significance of FLT3.

Every APL patient diagnosed in our institutions will follow our guidelines with respect to diagnosis procedures. Risk category will depend on white blood cell counts (WBC), where WBC >10000 will be considered high risk (HR) and <10000 WBC, low risk (LR).

Patients will receive induction with ATO plus ATRA daily until hematologic remission or for a maximum of 60 days, followed by ATO 5 days/week, 4 weeks on 4 weeks off, for a total of 4 courses and ATRA 2 weeks on and 2 weeks off for a total of 7 courses.

HR patients will receive 2-3 doses of IDA at the beginning of induction. Central nervous system prophylaxis is contemplated for HR pts or those who have SNC bleeding.

Molecular response will be evaluated at the end of consolidation by RQ-PCR. LR patients who achieve CMR will not need to repeat molecular evaluations but HR patients will need RQ-PCR evaluation every 3 months during the first year and every 6 months during the second year.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Signature of the form consent for participation in the study.
* Diagnosis of APL (either primary or secondary) according to the criteria of the World Health Organization (WHO), without prior treatment.
* Identification of the specific genetic alteration of APL by conventional karyotype, fluorescent in situ hybridization (FISH), reverse transcriptase polymerase chain reaction (RT-PCR or RQ-PCR). Identification of the transcript is recommended at the time of diagnosis isoforms: bcr1, bcr2, bcr3 essential to document the therapeutic response: Molecular remission

Exclusion Criteria:

* Presence of other concomitant active malignant tumors that require simultaneous treatment.
* Having received prior treatment for APL.
* Electrocardiogram abnormalities:

  1. Patients with a pre-existing diagnosis of Long QT Syndrome
  2. Patients with a baseline QTc of> 450msec. The Bazett formula should be used to measure the corrected QT interval (QT interval in msec divided by the square root of the RR interval in msec).
  3. Patients with a history or presence of significant ventricular or atrial tachyarrhythmia (Grade 3-4, CTCAE v5.2017).
  4. Patients with right bundle branch block plus left anterior hemiblock. Bifascicular blocks are excluded.
* ECOG score 4.
* Stage III-IV heart failure.
* Serum creatinine ≥ 2.5 mg / dL (≥ 250 μmol / L) unless due to APL.
* Bilirubin ≥ 2.5 mg / dL, alkaline phosphatase, GPT or GOT> 3 times the normal limit unless it is for APL.
* Severe psychiatric illness.
* Women who are pregnant or who have decided to continue breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with APL in first line treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate overall survival of patients diagnosed with APL and treated in first line with ATO/ATRA or ATO/ATRA/Idarubicin (IDA). | 36 months
  Evaluate overall survival of patients >/= 18 years old diagnosed with APL and treated in first line with ATO/ATRA or ATO/ATRA/Idarubicin (IDA) depending on risk category.
Evaluate event free survival of patients diagnosed with APL and treated in first line with ATO/ATRA or ATO/ATRA/Idarubicin (IDA). | 36 months
  Evaluate event free survival of patients >/= 18 years old diagnosed with APL and treated in first line with ATO/ATRA or ATO/ATRA/Idarubicin (IDA) depending on risk category.

SECONDARY OUTCOMES:
Evaluate complete molecular remission rate at the end of the consolidation treatment. | 36 months
Evaluate toxicity of the ATO/ATRA scheme (+/- IDA), measured according to type, frequency, severity and relation with the treatment of adverse events. | 36 months
Record early mortality (within 30 days of admission). | Within 30 days of admission
Evaluate whether the presence of mutated FLT3 has prognostic value in patients treated with ATRA/ATO. | 36 months
  The prognostic value will be analyzed by comparing rates of complete remission (CR), hematological relapse, molecular relapse, PFS and OS.

CONTACTS AND LOCATIONS:
Overall Officials: María José Mela Osorio, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda; Isolda Fernández, Dr., Study Chair — Grupo Argentino de Tratamiento de la Leucemia Aguda; Federico Sackmann, Dr., Principal Investigator — Grupo Argentino de Tratamiento de la Leucemia Aguda
Locations (6):
- Argentina (6):
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Instituto Privado de Hematologia y Hemoterapia, Paraná, Entre Ríos Province
  - Hospital Escuela de Agudos Dr. Ramón Madariaga, Posadas, Misiones Province
  - Hospital Descentralizado Dr. Guillermo Rawson, Rawson, San Juan Province
  - CEMIC, CABA
  - FUNDALEU, CABA

IPD SHARING:
Plan to Share IPD: Yes
Share study protocol
Supporting Information: Study Protocol
Time Frame: The data will become available on June 2021, and will remain available until the end of the clinical trial.